CLINICAL TRIAL: NCT01986166
Title: A Phase Ib, Open-Label, Dose-Escalation Study of the Safety, Tolerability, and Pharmacokinetics of MEHD7945A and Cobimetinib in Patients With Locally Advanced or Metastatic Solid Tumors With Mutant KRAS
Brief Title: A Study of MEHD7945A and Cobimetinib in Patients With Locally Advanced or Metastatic Cancers With Mutant KRAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29030; 2013-001910-14 (EudraCT Number)
Record Dates: First submitted 2013-11-01; First posted 2013-11-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — cobimetinib; MEHD7945A

ARMS (3):
- MEHD7945A + Cobimetinib - Stage 1 (Experimental): Patients will receive MEHD7945A 1100 milligrams (mg) intravenous (IV) infusion every 2 weeks (q2w) in combination with cobimetinib. Cobimetinib will be administered at a starting dose of 80 mg oral tablet q2w. Cobimetinib doses will be escalated to establish maximum tolerated dose (MTD) of MEHD7945A+cobimetinib combination for Stage 2.
  Interventions: Drug: Cobimetinib; Drug: MEHD7945A
- MEHD7945A + Cobimetinib - Stage 2 (CRC) (Experimental): CRC patients will receive MEHD7945A in combination with cobimetinib until disease progression or unacceptable toxicity. The doses and schedule of the combination treatment will be according to the MTD established in Stage 1.
  Interventions: Drug: Cobimetinib; Drug: MEHD7945A
- MEHD7945A + Cobimetinib - Stage 2 (NSCLC) (Experimental): NSCLC patients will receive MEHD7945A in combination with cobimetinib until disease progression or unacceptable toxicity. The doses and schedule of the combination treatment will be according to the MTD established in Stage 1.
  Interventions: Drug: Cobimetinib; Drug: MEHD7945A

INTERVENTIONS:
Drug: Cobimetinib — In Stage 1, cobimetinib will be administered at a starting dose of 80 mg q2w. The doses will be escalated to identify MTD. In Stage 2, participants will receive cobimetinib at the established MTD.
  Other Names: GDC-0973
Drug: MEHD7945A — MEHD7945A will be administered as IV infusion at a dose of 1100 mg q2w until disease progression or unacceptable toxicity.
  Other Names: Duligotuzumab

SUMMARY:
This open-label, multicenter, global Phase Ib study will evaluate the safety, tolerability and pharmacokinetics of intravenous (IV) dosing of MEHD7945A in combination with oral dosing of cobimetinib in patients with locally advanced or metastatic solid tumors that carry a Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) mutation and for which standard therapies do not exist, have proven ineffective or intolerable or are considered inappropriate. The study comprises a dose-escalation (Stage 1) and an indication-specific cohort expansion stage (Stage 2).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic solid KRAS-mutant tumors, for which standard therapies do not exist, have proven ineffective or intolerable or are considered inappropriate
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Evaluable disease or disease measurable per modified Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Consent to provide archival tumor tissue for biomarker testing
* Additionally, for patients who are considered for enrollment into the indication specific expansion cohorts in Stage 2, the current cancer must be either KRAS-mutant colorectal cancer (CRC) or KRAS-mutant non-small cell lung cancer (NSCLC)

Exclusion Criteria:

* History of prior significant toxicity from another MEK pathway inhibitor or combination of another MEK and epidermal growth factor receptor (EGFR) inhibitor requiring discontinuation of treatment
* Previous treatment with a combination of a MEK inhibitor with an EGFR inhibitor (applies only to the indication specific expansion cohorts in Stage 2)
* Allergy or hypersensitivity to components of the cobimetinib formulations
* History of severe (Grade 3 or 4) allergic or hypersensitivity reaction to therapeutic antibodies that required discontinuation of therapy
* History of interstitial lung disease (ILD)
* Known severe ulcer disease
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, central serous chorioetinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration

Patients will be excluded if they currently have either of the following conditions which have been identified as risk factors for CSCR:

* Uncontrolled glaucoma with intraocular pressure greater than (>) 21 millimeters of mercury (mm Hg)
* Grade greater than equal to (>=) 3 hypertriglyceridemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with adverse events | up to approximately 2 years
Percentage of patients with anti-MEHD7945A antibodies | up to approximately 2 years
Percentage of patients with dose-limiting toxicities (DLTs) | 28 days

SECONDARY OUTCOMES:
Percentage of patients with fluorodeoxyglucose positron emission tomography (PET) response, defined as a >=20% decrease in fluorodeoxyglucose uptake by PET | Baseline, Day 15 of Cycle 1 (cycle length=28 days)
MEHD7945A maximum serum concentrations (Cmax) | Pre-dose (0 hour) on Days 1, 15 and 0.5 hour post-infusion (infusion duration=1.5 hour) on Days 1, 15 of Cycles 1, 2 and pre-dose (0 hour) and 0.5 hour post-infusion (infusion duration=1 hour) on Day 15 of Cycle 4 (up to 14 weeks) (cycle length=28 days)
MEHD7945A minimum serum concentrations (Cmin) | Pre-dose (0 hour) on Days 1, 15 of Cycles 1, 2 and pre-dose (0 hour) on Day 15 of Cycle 4 (up to 14 weeks) (cycle length=28 days)
Cobimetinib area under the concentration-time curve (AUC) | Pre-dose (0 hour), 1, 2, 4 hour post-infusion (infusion duration=1.5 hour) on Cycle 1 Days 1 & 15 and Cycle 4 Day 15, 6 & 24 hours post-infusion on Cycle 1 Day 15, 6 hour post-infusion on Cycle 4 Day 15 (up to 14 weeks) (cycle length=28 days)
Cobimetinib maximum plasma concentrations (Cmax) | Pre-dose (0 hour), 1, 2, 4 hour post-infusion (infusion duration=1.5 hour) on Cycle 1 Days 1 & 15 and Cycle 4 Day 15, 6 & 24 hours post-infusion on Cycle 1 Day 15, 6 hour post-infusion on Cycle 4 Day 15 (up to 14 weeks) (cycle length=28 days)
Time to maximum cobimetinib plasma concentration (tmax) | Pre-dose (0 hour), 1, 2, 4 hour post-infusion (infusion duration=1.5 hour) on Cycle 1 Days 1 & 15 and Cycle 4 Day 15, 6 & 24 hours post-infusion on Cycle 1 Day 15, 6 hour post-infusion on Cycle 4 Day 15 (up to 14 weeks) (cycle length=28 days)
Percentage of patients with objective response | Baseline, Days 22 of Cycle 2 and Day 25 of Cycle 4 and then every 8 weeks throughout the duration of the study (up to approximately 2 years) (cycle length=28 days)
Duration of objective response | Baseline, Day 22 of Cycle 2 and Day 25 of Cycle 4 and then every 8 weeks throughout the duration of the study (up to approximately 2 years) (cycle length=28 days)
Progression-free survival | Baseline, Day 22 of Cycle 2 and Day 25 of Cycle 4 and then every 8 weeks throughout the duration of the study (up to approximately 2 years) (cycle length=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (9):
- United States (6):
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Detroit, Michigan
  - Nashville, Tennessee
  - Dallas, Texas
- Spain (3):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia

REFERENCES:
- [Derived] Lieu CH, Hidalgo M, Berlin JD, Ko AH, Cervantes A, LoRusso P, Gerber DE, Eder JP, Eckhardt SG, Kapp AV, Tsuhako A, McCall B, Pirzkall A, Uyei A, Tabernero J. A Phase Ib Dose-Escalation Study of the Safety, Tolerability, and Pharmacokinetics of Cobimetinib and Duligotuzumab in Patients with Previously Treated Locally Advanced or Metastatic Cancers with Mutant KRAS. Oncologist. 2017 Sep;22(9):1024-e89. doi: 10.1634/theoncologist.2017-0175. Epub 2017 Jun 7. PMID 28592615